CLINICAL TRIAL: NCT01316809
Title: Phase I Trial of AZD8055, An Oral MTOR Kinase Inhibitor, for Adults With Recurrent Gliomas
Brief Title: AZD8055 for Adults With Recurrent Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110122; 11-C-0122
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2016-04-14

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Malignant Glioma; Brainstem Glioma
Keywords: Brain; Tumor; Recurrent; Surgery; Radiation; Glioma; Brain Tumor; Glioblastoma Multiforme; Astrocytoma; Brainstem Glioma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Neoplasms; Recurrence; Brain Neoplasms | interventions — (5-(2,4-bis((3S)-3-methylmorpholin-4-yl)pyrido(2,3-d)pyrimidin-7-yl)-2-methoxyphenyl)methanol

ARMS (2):
- A (Experimental): Surgical arm
  Interventions: Drug: AZD8055
- B (Experimental): Non-surgical arm
  Interventions: Drug: AZD8055

INTERVENTIONS:
Drug: AZD8055 — Patients will start at 120 mg once daily

SUMMARY:
Background:

- AZD8055 is an experimental cancer treatment drug that works by inhibiting a protein called mTOR, which is known to promote tumor cell and blood vessel growth and to control tumor s energy and nutrient levels. AZD8055 is the first drug that inhibits both types of mTOR protein and is expected to be more effective than prior mTOR inhibitors. However, more research is needed to determine its safety and effectiveness in treating brain tumors known as gliomas that have not responded to standard treatments.

Objectives:

- To evaluate the safety and effectiveness of AZD8055 in individuals with gliomas that have not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with gliomas that have not responded to standard chemotherapy, surgery, or radiation.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, and tumor imaging studies.
* Participants will be separated into two treatment groups: one group that will receive surgery to remove the glioma and one that will not have surgical treatment.
* Participants in the nonsurgical treatment group will take AZD8055 by mouth daily for a 42-day cycle of treatment. Participants will keep a diary to record doses and keep track of any side effects.
* Participants in the surgical treatment group will take AZD8055 by mouth daily for 7 days, and then will have tumor removal surgery. At least 3 weeks after surgery, participants will resume doses of AZD8055 and will continue to take the drug for as long as the tumor does not recur.
* During treatment, participants will have regular visits to the clinical center, involving frequent blood and urine tests and other examinations to monitor the effects of treatment. Participants will have imaging studies to study the cancer's response to the treatment.
* Participants will continue to have cycles of treatment for as long as the treatment continues to be effective and the side effects are not severe enough to stop participation in the study....

DETAILED DESCRIPTION:
Background:

* Recurrent glioma patients have very limited treatment options. A significant percentage of gliomas have increased activity of the PI3K/Akt/mTOR pathway, mostly due to loss of PTEN.
* AZD8055 is a first in-class inhibitor of the kinase activity of mTOR, specifically inhibiting both mTORC1 and mTORC2 complexes. Preclinical data generated in the Neuro-Oncology Branch Laboratory of Dr. Howard Fine demonstrated that AZD8055 has significant anti-glioma activity in vivo and in vitro.

Objectives:

* To establish the maximally tolerated dose (MTD) of continuous once daily AZD8055 in patients with recurrent malignant gliomas not on enzyme-inducing anti-epileptic drugs (EIAED).
* To generate pharmacokinetic data on continuous once daily AZD8055 dosing.

Eligibility:

-Patients with histologically proven glioma are eligible for this study. Patients should have failed prior standard treatment with radiotherapy.

Design:

* This study will accrue up to 24 evaluable patients (non-surgical arm). Cohorts of 3 or 6 patients will receive continuous AZD8055 once daily orally for 42 days. The MTD will be based on the tolerability observed during the first 6 weeks of treatment only. Up to three patients may be enrolled simultaneously at each dose level. The dose of AZD8055 can be progressively escalated if only 0/3 or 1/6 patients experience a dose limiting toxicity at the prior dose level.
* A subset of patients in whom tumor re-resection is considered standard of care will receive 1-week treatment with AZD8055 and then undergo resection. Patients will be treated at the highest dose level shown to be safe at the time of enrollment. Once patients recover from surgery, they will restart treatment with AZD8055 and stay on treatment as long as there is no tumor progression or protocol-mandated removal criteria. Management of toxicity will be the same as non-surgical patients receiving their second and subsequent cycles of therapy as delineated in the protocol. Up to 12 patients will enter the surgical arm of this trial.
* The accrual ceiling will be open to 42 patients to factor in replacing those who come off

treatment prior to cycle 1.

-At the end of Cycle 1, patients in both treatment arms (surgical and non-surgical) may choose to continue to receive AZD8055 until disease progression or until they experience unmanageable drug related toxicity, as long as they are continuing to derive clinical benefit and do not fulfill any of the criteria for removal from protocol therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically proven malignant primary gliomas who have progressive disease after radiotherapy will be eligible for this protocol. These include glioblastoma (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), and malignant glioma/astrocytoma NOS. Additionally, patients with progressive low-grade gliomas and patients with infiltrative brainstem gliomas, diagnosed radiographically rather than by biopsy, will be eligible.
* Patients must have an MRI scan performed within 14 days prior to registration and on a fixed dose of steroids for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MRI is required.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible for the non-surgical arm as long as all of the following conditions apply:

  1. Patients will be eligible four weeks after surgery if they have recovered from the effects of surgery.
  2. Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease postoperatively, an MRI should be done:

     * no later than 96 hours in the immediate post-operative period or
     * at least 4 weeks post-operatively, and
     * within 14 days of registration, and
     * on a stable steroid dosage for at least 5 days.

If the 96 hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI is required on a stable steroid dosage for at least 5 days.

* Patients must have failed prior radiation therapy.
* All patients or their previously designated DPA (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must be greater than or equal to 18 years old, and must have a life expectancy > 8 weeks.
* Patients must have a Karnofsky performance status of greater than or equal to 60.
* Patients must be at least 4 weeks from radiation therapy. Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide, 3 weeks from procarbazine, 2 weeks from vincristine and 2 weeks from last bevacizumab administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen) including investigative agents. With the exception of alopecia, all toxicities from prior therapies should be resolved to CTCAE less than or equal to grade 1.
* Patients must have adequate bone marrow function (WBC greater than or equal to 3,000/microL, ANC greater than or equal to 1,500/mm(3), platelet count of greater than or equal to 100,000/mm(3), and hemoglobin greater than or equal to 9 gm/dl), adequate liver function (AST, ALT and alkaline phosphatase 2.5 less than or equal to ULN and bilirubin less than or equal to 1.5 times ULN), and adequate renal function (creatinine less than or equal to 1.5 times ULN and/or creatinine clearance greater than or equal to 50 cc/min calculated by Cockcroft-Gault) before starting therapy. Patients must also have serum potassium greater than or equal to 3.5 mmol/L, magnesium greater than or equal to 0.75 mmol/L and calcium levels within normal levels; supplementation is allowed. In cases where the serum calcium is below the normal range, 2 options would be available: 1) the calcium adjusted for albumin is to be obtained and substituted for the measured serum value. Exclusion is to then be based on the adjusted for albumin values falling below the normal limit. 2) Determine the ionized calcium levels. Exclusion is then to be based if these ionized calcium levels are out of normal range despite supplementation. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
* Patients must either not be receiving steroids, or be on a stable dose of steroids for at least five days prior to registration.
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.
* Male patients should be willing to use barrier contraception (condoms).
* Female patients should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* A 12 lead electrocardiogram (ECG) to be performed within 2 weeks of trial entry with QTc less than or equal to 470 msec.
* Patients must have normal left ventricular ejection fraction (LVEF greater than or equal to 55% or normal by NIH Clinical Center criteria).

EXCLUSION CRITERIA:

* Patients who, in the view of the treating physician, have significant active hepatic, renal, pulmonary or psychiatric diseases are ineligible.
* Prior treatment with AZD8055 or AZD2014.
* History of hypersensitivity to active or excipients of AZD8055 or drugs with a similar chemical structure or class to AZD8055.
* Clinically significant cardiovascular event (e.g. myocardial infarction, angina pectoris, coronary artery bypass graft, angioplasty, vascular stent, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease greater than or equal to 2 within 6 months before entry; or presence of cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
* Hemorrhagic or ischemic stroke, including transient ischemic attacks and other central nervous system bleeding in the preceding 6 months that were not related to glioma surgery. History of prior intratumoral bleeding is not an exclusion criteria; patients with history of prior intratumoral bleeding, however, need to undergo a non-contrast head CT to exclude acute blood.
* Ventricular arrhythmias requiring continuous therapy or asymptomatic sustained ventricular tachycardia within 12 months before study entry. Atrial fibrillation, controlled on medication is not excluded. Patients with significant ECG abnormalities such as complete left bundle block and third degree heart block are not eligible.
* QTc prolongation with other medications that required discontinuation of that medication.
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.
* QTc with Bazett s correction that is unmeasurable, or >470 msec on screening ECG. (Note: If a subject has a QTc interval >470 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be less than or equal to 470 msec in order for the subject to be eligible for the study. Patients who are receiving a drug that has a risk of QTc prolongation are excluded if QTc is greater than or equal to 460 msec.
* Any concurrent medication that may cause QTc prolongation or induce Torsades de Pointes Drugs, that in the investigator s opinion cannot be discontinued are allowed; however, must be monitored closely.
* Concomitant medications that are moderate or potent inducers of CYP3A4 or CYP2C8 function (with the exception of dexamethasone) are not permitted within the specified wash-out periods prior to or during treatment with AZD8055.
* Patients with uncontrolled hypercholesterolemia or hypertriglyceridemia (fasting state) despite lipid-lowering therapy.
* Patients with manifest diabetes mellitus type 1 and patients with uncontrolled diabetes mellitus type 2 or corticosteroid-induced hyperglycemia despite optimal therapy.
* Refractory nausea and vomiting or significant gastrointestinal impairment, as judged by the investigator, that would significantly affect the absorption of AZD8055, including the ability to swallow the tablet whole.
* Patients known to have active hepatitis B or C or HIV on anti-retrovirals (testing is not required for entry on study).
* Other concomitant anti-cancer therapy except corticosteroids.
* Patients with a peripheral neuropathy CTCAE > 1 in the prior 4 weeks or active muscle diseases (including dermatomyositis, polymyositis, inclusion body myositis, muscular dystrophy and metabolic myopathy) or family history of myopathy.
* Patients with pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi syndrome or renal tubular acidosis.
* Evidence of active infection or active bleeding diatheses.
* Patients with an abnormal LVEF on echocardiogram at baseline.
* Women who are currently pregnant or breast feeding.
* Patients known to have a malignancy (other than their malignant glioma) that has required treatment in the last 12 months and/or is expected to require treatment in the next 12 months (except for non-melanoma skin cancer, carcinoma in situ in the cervix or ductal carcinoma in situ).
* Major surgery within 4 weeks or incompletely healed surgical incision before starting therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-03-04; Primary Completion 2014-04-14 (Actual); Study Completion 2016-04-04 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) of AZD8055 on a continuous once daily schedule in patients with recurrent gliomas not on enzyme-inducing anti-epileptic drugs (EIAED). | 2 years
Generate pharmacokinetic data of AZD8055 on a continuous once daily schedule | 2 years

SECONDARY OUTCOMES:
To obtain exploratory information about the antitumor activity of AZD8055. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] FRANKEL SA, GERMAN WJ. Glioblastoma multiforme; review of 219 cases with regard to natural history, pathology, diagnostic methods, and treatment. J Neurosurg. 1958 Sep;15(5):489-503. doi: 10.3171/jns.1958.15.5.0489. No abstract available. PMID 13576192
- [Background] Bloom HJ. Combined modality therapy for intracranial tumors. Cancer. 1975 Jan;35(1):111-20. doi: 10.1002/1097-0142(197501)35:13.0.co;2-#. PMID 162849
- [Background] Salazar OM, Rubin P, Feldstein ML, Pizzutiello R. High dose radiation therapy in the treatment of malignant gliomas: final report. Int J Radiat Oncol Biol Phys. 1979 Oct;5(10):1733-40. doi: 10.1016/0360-3016(79)90554-6. No abstract available. PMID 231023